CLINICAL TRIAL: NCT06242704
Title: Train Your Brain 2.0: Improving Memory and Decision Making to Improve Outcomes Among Youth - A Randomized Controlled Trial
Brief Title: Train Your Brain 2.0 - Improving Memory and Decision Making Among Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Julia Felton, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B11256
Record Dates: First submitted 2024-01-16; First posted 2024-02-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Behavior, Health
Keywords: delay discounting; computer-based intervention; executive functioning; substance use; working memory
MeSH Terms: conditions — Health Behavior; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working Memory Training (Experimental): The intervention is a computer-based training aimed at improving working memory in order to decrease delay discounting. Active training sessions include: Sequenced Recall of Digits - Auditory, Sequenced Reverse Recall of Digits - Auditory, Sequenced Recall of Digits - Visual, Sequenced Reverse Recall of Digits - Visual, Sequenced Recall of Words - Auditory, Sequenced Recall of Words - Visual, Sequenced Reverse Recall of Words - Auditory, Sequenced Reverse Recall of Words - Visual. Participants will complete at least 10 sessions with each session taking approximately 30 minutes to complete.
  Interventions: Behavioral: Working Memory Training
- Working Memory (Active Comparator): The comparison control condition is a multi-session control computer training condition that is designed to not engage working memory during computer-based engagement sessions: Sequenced Recall of Digits - Auditory, Sequenced Reverse Recall of Digits - Auditory, Sequenced Recall of Digits - Visual, Sequenced Reverse Recall of Digits - Visual, Sequenced Recall of Words - Auditory, Sequenced Recall of Words - Visual, Sequenced Reverse Recall of Words - Auditory, Sequenced Reverse Recall of Words - Visual. Participants will complete at least 10 sessions with each session taking approximately 30 minutes to complete.
  Interventions: Behavioral: Working Memory

INTERVENTIONS:
Behavioral: Working Memory Training — A multi-session computer-based working memory training program to improve delay discounting and prevent substance use among at-risk adolescents in a traditionally underserved area.
  Arms: Working Memory Training
Behavioral: Working Memory — A multi-session control computer training condition that is designed to not engage working memory among at-risk adolescents in a traditionally underserved area.
  Arms: Working Memory

SUMMARY:
The goal of this clinical trial is to deliver a computer-based working memory training program to improve delay discounting (DD) and prevent substance misuse among at-risk adolescents in a traditionally underserved area. Results from the study will inform future substance use prevention efforts targeted at youth exposed to adverse childhood experiences. Findings will also refine future models of intervention delivery in traditionally underserved communities.

The main aims of the project are are:

1) To examine to examine changes in hypothesized mechanisms of substance use initiation and escalation, and 2) to assess whether changes in DD are a mechanism for reducing substance misuse during early adolescence. The investigators will evaluate whether changes in DD following active treatment predict substance use outcomes over the three-month follow-up period.

DETAILED DESCRIPTION:
Youth exposed to early childhood adversity are at increased risk for engaging in problematic substance use, leading to myriad negative health outcomes, including HIV exposure, injury, and impaired driving. Adolescents from low-resource communities evidence elevated rates of exposure to adverse childhood experiences, yet have limited access to evidence-based preventative interventions. Thus, there is a critical need for services that can feasibly target specific mechanisms linking early adversity to the onset and escalation of substance use in traditionally underserved communities.

One such target is delay discounting (DD), the tendency to select small, immediately available rewards relative to larger, delayed, rewards. DD has been linked to early substance use initiation and more frequent and severe use across adolescence. Moreover, youth exposed to early childhood adversity evidence more problematic levels of DD, indicating that DD may be a pathway by which early trauma exposure leads to drug and alcohol use.

Research from the investigative team suggests that computer-based interventions targeting proximal cognitive skills, specifically working memory, can improve rates of DD. Moreover, computerized interventions are highly transportable and scalable, making them ideal for dissemination in low-resource communities. The current project proposes to pilot a computer-based working memory (WM) training program to improve DD and prevent substance use among at-risk adolescents in a traditionally underserved area.

ELIGIBILITY:
Adolescent Inclusion Criteria:

1. Between the ages of 11 and 15 and have a parent/guardian willing to provide consent for their participation
2. Proficient in English
3. Willing to commit to participate in computer-based trainings over the course of 5-8 weeks (duration dependent on site)
4. Access to internet services, cell phone, and/or email
5. Willing to receive/send study-related text messages

Adolescent Exclusion Criteria:

1. Self-disclosure or identification with psychological disturbance, suicidality, or evidence of active suicide ideation
2. Self-disclosure of current substance use disorder

Parent Inclusion Criteria:

1. Provide consent for child's participation in study
2. Proficient in English
3. Access to internet services, cell phone, and/or email
4. Willing to receive/send study-related text messages

Parent Exclusion Criteria:

1. Self-disclosure or identification with psychosis, suicidality, or evidence of active suicide ideation
2. Self-disclosure of current substance use disorder

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Monetary Choice Questionnaire | Baseline, 2 Weeks, 3 Months
  The Monetary Choice Questionnaire (MCQ) is a measure of delay discounting (DD). Participants will be presented with two choices, one with a small, immediate monetary reward and the other with a larger, delayed monetary reward. They will be required to choose one of those rewards and their responses will be scored using reference discounting curves. A calculated score that places participants on steeper curves indicates higher levels of impulsivity and higher rates of DD. Scores are not bounded with a minimum and maximum value, but higher scores indicate worse outcomes and demonstrate the participant's preference to gain smaller rewards immediately over larger rewards with a time delay.

SECONDARY OUTCOMES:
Change in Consideration of Future Consequences Scale | Baseline, 2 Weeks, 3 Months
  The Consideration of Future Consequences Scale1 (CFCS-14) is a 14-item self-report questionnaire that assesses active consideration of longer-term implications of an individual's actions. Lower scores on the CFCS-14 are associated with a greater focus on immediate needs and have been found to be associated with less engagement in health behaviors and greater substance use. Individual items are rated on a scale from 1 to 7 with total scores range from 14-98. The measure has been used extensively among adult samples and demonstrates strong reliability and validity. Research suggests modest but significant correlations with the Monetary Choice Questionnaire (MCQ). Change in CFCS-14 score is measured by comparing baseline scores with scores at the post-intervention assessment with higher scores reflecting greater increases in future thinking.
Change in Digit Span | Baseline, 2 Weeks, 3 Months
  The Digit Span Task is a measure of memory. Participants are presented with digit sequences of increasing length and are required to recall them either in forward order (Digit Span Forward) or in reverse order (Digit Span Backward). Digit Span Forward is a measure of immediate memory and Digit Span Backward is a measure of working memory. Participants will move up or down levels based on correct or incorrect recall of sequences, respectively. Moving up a level will increase the sequence length while moving down a level will decrease the sequence length. Standardized scores range from 0 to 20. Higher scores in this task indicate better performance over 14 trials. Computerized memory tasks such as this have demonstrated increased reliability in short-term memory assessments.
Change in Stop Signal Task | Baseline, 2 Weeks, 3 Months
  The Stop Signal Task (SST) is a measure of response inhibition. Participants are first presented with either a left pointing arrow or a right pointing arrow. They are required to select the left arrow button upon seeing a left pointing arrow and the right arrow button upon seeing the right pointing arrow. After 16 trials, a second component is added to the task. Participants will continue to select left or right arrow buttons, but once they are presented with an auditory cue (a beep), they need to withhold their response. The delay in presenting the auditory cue after the arrow is shown (Stop Signal Delay; SSD) will become longer or smaller based on participant performance. The stop signal response time (SSRT) gives an estimate of the time it takes for a response to be stopped upon hearing the cue. Longer SSRT generally indicates poor performance on the SST. Standardized scores range from 0 to 100 with greater scores representing better task performance.
Changes in Letter Number Sequencing Test | Baseline, 2 Weeks, 3 Months
  Letter Number Sequencing (LNS) is a measure of working memory. This test has two parts to it: the forward test and the reordered test. In the forward test, the participant is visually presented with a list of scrambled letters and numbers that they must type into a text box in the same alphabetical and numeric order that was presented. In the reordered test, the participant is visually presented with a list of scrambled letters and numbers that they must type into a text box with numbers listed first in ascending order and letters listed second in alphabetical order. The length of the target string increases over time until the participant is no longer able to correctly sequence three letter/ number stems in a row. The investigators will use a computerized version of the LNS test. Higher scores in this test indicate better outcomes with standardized scores ranging from 0 to 20.
Change in Alcohol Effect Expectancies (Breif) | Baseline, 2 Weeks, 3 Months
  The Alcohol Expectancy Questionnaire-Brief (AEQ-B) is a self-report questionnaire that tap youths' perception of positive and negative outcomes related to using alcohol. Because this intervention is designed to orient youth towards longer-term (rather than immediate) rewards, the investigators expect to see significant decreases in positive expectancies of alcohol use and an increase in negative expectations. The AEQ has been found to be reliable and valid indicators of adolescents' perceptions of use. Seven items on the questionnaire are rated on a 1 to 5 scale, with higher scores generally indicating worse outcomes. Scores range from 7 to 35.
Change in Marijuana Effect Expectancies | Baseline, 2 Weeks, 3 Months
  The Marijuana Effect Expectancy Questionnaire-Brief (MEEQ-B) is a self-report questionnaire that tap youths' perception of positive and negative outcomes related to using marijuana. Because this intervention is designed to orient youth towards longer-term (rather than immediate) rewards, the investigators expect to see significant decreases in positive expectancies of marijuana use and an increase in negative expectations. The MEEQ has been found to be reliable and valid indicators of adolescents' perceptions of use. Six items on the questionnaire are rated on a 1 to 5 scale, with higher scores generally indicating worse outcomes. Scores range from 6 to 30.
Change in Youth Risk Behavior Survey | Baseline, 2 Weeks, 3 Months
  The Youth Risk Behavior Survey (YRBS) is a self-report measure of the prevalence of real world risk behaviors, including compromised safety behaviors (e.g. not wearing a seat belt), substance use, risky sexual practices, and delinquent behaviors (e.g. gambling, theft). Because substance use has been associated with problematic behaviors more broadly, the YRBS will allow us to tap engagement in a variety of related risky behaviors. Consistent with previous research, the investigators will create an aggregate of substance use and risk behaviors as an index of risky behaviors. Composite scores such as these have demonstrated adequate psychometric properties. There are 71 items on the scale that will be analyzed at the item level. Most items on the survey are reported on a 0 to 5 scale, with the score of 5 indicating riskier behavior.
Change in Balloon Analogue Risk Test - Youth | Baseline, 2 Weeks, 3 Months
  The Balloon Analogue Risk Test - Youth (BART-Y) is a measure of risk aversion. It requires participants to choose between continuing to pump a balloon or collecting the winnings they already earned from pumping the balloon before. Participants will earn money for every successful pump where the balloon remains unexploded. If the balloon explodes before they collect their winnings, they will lose all the money they could have collected from the given balloon. Participants are given 30 balloons in this task. The average number of pumps for the unexploded balloons is calculated at the end, where a higher number of average pumps indicates worse outcomes (greater risk seeking behavior and lower risk aversion). Scores range from 0 to the maximum number of pumps before the balloon explodes which varies across the task.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Freedom Schools Collaborative, Flint, Michigan
  - Ernest T. Ford Recreation Center, Highland Park, Michigan